CLINICAL TRIAL: NCT05736445
Title: Evaluating Student Wellness Using a Blended Approach of the Roadmap mHealth App Plus Wellness Coaching
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sung Won Choi, Edith S Briskin and Shirley K Schlafer Foundation Research Professor of Pediatrics, Professor of Pediatrics, University of Michigan Medical School, University of Michigan
Other Study IDs: HUM00223936
Record Dates: First submitted 2023-01-26; First posted 2023-02-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Students at the University of Michigan: Students enrolled in the Winter 2023 academic semester at the University of Michigan
  Interventions: Behavioral: Wellness coaching plus app use

INTERVENTIONS:
Behavioral: Wellness coaching plus app use — Participants will participate in wellness coaching and interact with apps on their smartphones

SUMMARY:
In this pilot study, the investigators plan to examine how the combination of wellness coaching and a mobile health app that promotes positive psychology activities can improve the overall well-being of college students. With these tools, the investigators hope to better understand the relationship between digital intervention and coaching and determine how it may improve the mental health of students. The study team also hopes to investigate how mental health can impact academic performance.

DETAILED DESCRIPTION:
Students seeking wellness coaching will have the option to participate in this study. The study will ask participants to:

1. Complete as many sessions of individual wellness coaching as they see fit
2. Install and interact with the Fitbit and Roadmap 2.0 apps on their smartphone
3. Complete longitudinal surveys at baseline, month 1, month 2, and end of study
4. Complete an exit interview at the end of the study
5. Allow the study team to access academic records (optional)

The investigators plan to evaluate the app + coaching influence on mental health outcomes and to determine what can be learned to improve its design for a future, full-scale study, if there is evidence of adoption and sustainability from this pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. University of Michigan students aged 18 years or older.
2. Students must either be coming to campus for the academic year or taking classes online for the academic year.
3. For those completing school online, must be able to provide a mailing address within the United States where they can receive study tools and be mailed study materials
4. Possess a smartphone (Apple or Android).
5. Ability to understand and demonstrate willingness to remotely sign a written informed consent.

Exclusion Criteria:

1. People who are not enrolled in classes at the University of Michigan for the Winter 2023 term.
2. Unwilling or unable to comply with the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Students enrolled at the University of Michigan
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Wellness Coaching + App Use | 9 months
  To assess the primary endpoint, the investigators will evaluate participants' opinions about the uptake of Roadmap + Wellness Coaching through semi-structured qualitative interviews. The investigators will ask questions related to the feasibility and acceptability of the: 1) Roadmap 2.0 app; 2) Fitbit device; 3) completing assessments (through the app); and 4) wellness coaching. The investigators expect the net favorability (agree + totally agree) of all four components will be >50% based on answering questions on a scale of totally disagree, disagree, neutral, agree, and totally agree to be considered feasible and acceptable to participate in.

SECONDARY OUTCOMES:
Survey Completion | 7 months
  Assess survey completion rate, estimating 50% of participants will complete the surveys at all four time points

CONTACTS AND LOCATIONS:
Overall Officials: Sung Won Choi, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States